CLINICAL TRIAL: NCT00001506
Title: Evaluation and Treatment of Subjects With Dermatologic Diseases
Brief Title: Evaluation and Treatment of Patients With Dermatologic Diseases
Status: Completed | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960102; 96-AR-0102; NCT00019149 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Dermatologic Diseases; Systemic Diseases With Cutaneous Manifestations
Keywords: Training; Standard Therapy; Standard Tests; Natural History; Consultation
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: With dermatologic diseases and systemic diseases with cutaneous manifestations

SUMMARY:
This is a training, natural history of disease, and screening protocol for the evaluation, treatment and follow-up of patients with dermatologic diseases and systemic diseases with cutaneous manifestations. Patients enrolled in this protocol will be evaluated and treated according to generally available, standard procedures and therapeutic modalities. Samples of blood and skin will be studied by routine and specialized investigative methods to establish these patients' diagnosis, response to treatment, and/or disease progression.

DETAILED DESCRIPTION:
Background

This is a training, natural history of disease, and screening protocol for the evaluation, treatment and follow-up of patients with dermatologic diseases and systemic diseases with cutaneous manifestations. This protocol was developed to allow subject enrollment for teaching purposes and to allow for second opinions regarding relatively complicated patients, and to allow for evaluation of non-invasive tools for the diagnosis and monitoring of cutaneous manifestations. This protocol promotes a critical link between the NCI, CCR Dermatology Branch and the local and national extramural medical communities.

Objectives:

* To provide clinical material to fulfill the educational mission of the Dermatology Branch.
* To learn about the natural history of selected dermatologic diseases.

Eligibility:

All subjects regardless of age, gender, or racial/ethnic group with dermatologic disease or systemic disease with cutaneous manifestations.

Design:

Patients enrolled in this protocol will be evaluated and treated according to generally available, standard procedures and therapeutic modalities. Samples of blood and skin will be studied by routine and specialized investigative methods to establish these patients diagnosis, response to treatment, and/or disease progression. Non-invasive tools may be used as part of the examination and assessment of cutaneous manifestations of disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients of any age (only viable neonates will enroll in the study), of both genders, and all racial/ethnic groups with dermatologic diseases or systemic diseases with cutaneous manifestations that will help the Branch fulfill the objectives.

Women who are pregnant or lactating, will only undergo tests and procedures, and/or receive medications for which data exists proving minimal risk to the fetus and/or child.

Patients must have a referring physician who will continue to assume primary medical responsibility of care for the patient during and after enrollment in this protocol.

EXCLUSION CRITERIA:

Any participant who, in the investigator s opinion, would be unable to comply with study requirements or for whom participation may pose a greater medical risk.

Ages: 1 Day to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with dermatologic diseases and systemic diseases with cutaneous manifestations
Sampling Method: Non-Probability Sample
Enrollment: 453 (Actual)
Dates: Start 1996-08-22 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Provide clinical material | Ongoing
  Provide clinical material
Natural history of selected dermatologic diseases | Ongoing
  Natural history of selected dermatologic diseases

CONTACTS AND LOCATIONS:
Overall Officials: Edward W Cowen, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Protocol is silent on individual participant data (IPD) sharing plan.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1996-AR-0102.html